CLINICAL TRIAL: NCT04699266
Title: Clinical Investigation of the Multifocal Intraocular Lens (IOL) POD F GF in Cataracteous Eyes
Brief Title: Clinical Investigation of the Multifocal IOL POD F GF in Cataracteous Eyes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beaver-Visitec International, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PHY2002
Record Dates: First submitted 2020-11-16; First posted 2021-01-07 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Cataract; Lens Opacities; Presbyopia
Keywords: Intraocular lens; Trifocal
MeSH Terms: conditions — Cataract; Presbyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: POD F GF IOL Implantation (Experimental): Experimental: POD F GF IOL Implantation experimental Multi-center, single-arm, non-masked study Mono- or bilateral implantation of trifocal intraocular lenses POD F GF
  Interventions: Device: Assigned Intervention (POD F GF)

INTERVENTIONS:
Device: Assigned Intervention (POD F GF) — The investigational lens (POD F GF )will be implanted to both eyes in subjects with bilateral cataract. Registration of patients and the implantation of the investigational lens (POD F GF) will be conducted in consideration of securing 44 eyes in 22 subjects as the analysis subjects

SUMMARY:
To evaluate effectiveness and safety of the POD F GF Intraocular Lens (IOL) when implanted to replace the natural lens following cataract removal

DETAILED DESCRIPTION:
Since the investigational lens, like conventional IOLs, is a posterior chamber lens which is widely implanted following cataract extraction, phacoemulsification is adopted. To assess the binocular vision, the investigational lens will be bilaterally implanted. Considering the safety of the study subjects, the time of implant to the remaining eye (2nd eye) will be decided based on the results of the 1st implant.

ELIGIBILITY:
Inclusion Criteria:

1. Adults, 20 years of age or older at the time of informed consent, of either gender, diagnosed with bilateral cataracts;
2. Able to comprehend and sign a statement of informed consent;
3. Willing and able to complete all required postoperative visits;
4. Calculated lens power within the available range;
5. Planned cataract removal by phacoemulsification;
6. Potential postoperative BCDVA of 0.5 decimal or better in both eyes;
7. Subject with preoperative astigmatism < 1.0 D
8. Clear intraocular media other than cataract in both eyes;
9. The subject must be able to undergo second eye surgery within 30 days of the first eye surgery.

[Justification for the inclusion criteria]

1. and 5: Cataract extraction is the indication of the clinical study.
2. and 3: One of GCP requirements 4: Essential condition for implant of the investigational lens. 6, 7, 8 and 9: Conditions to minimize the potential non-IOL factors which may affect the visual acuity data

Exclusion Criteria:

[Exclusion Criteria Prior to Surgery] The patient who meets any criteria specified in the following 1) through 22).

1. Irregular corneal aberration that affects postoperative visual function as demonstrated by corneal topography;
2. Inflammation or edema (swelling) of the cornea affecting post-operative visual acuity;
3. Subjects with diagnosed degenerative visual disorders (e.g. macular degeneration or other retinal disorders) that are predicted to cause future acuity losses to a level worse than 0.5 decimal for BCDVA;
4. Subjects who may be expected to require ocular surgery (other than blepharo-surgery, laser surgery of fundus and YAG capsulotomy) during the study;
5. Previous refractive surgery;
6. Amblyopia;
7. Clinically severe corneal dystrophy (eg., epithelial, stromal, or endothelial dystrophy), keratitis, keratoconjunctivitis, keratouveitis, keratopathy, or kerectasia;
8. Diabetic retinopathy;
9. Extremely shallow anterior chamber, not due to swollen cataract;
10. Microphthalmos;
11. Current or previous retinal detachment;
12. Previous corneal transplant;
13. Recurrent severe anterior or posterior segment inflammation of unknown etiology;
14. Rubella or traumatic cataract;
15. Iris neovascularization;
16. Glaucoma or ocular hypertension;
17. Aniridia;
18. Optic nerve atrophy;
19. Planned clear lensectomy (no lens opacity)
20. Pregnancy, lactating or possible pregnant;
21. Participation in any clinical study (drug or device) within 3 months prior to participating this study, planned participation another clinical study during this study, or currently participating in another study.
22. Disqualified by the investigator or the sub-investigator because of physical or ophthalmic diseases.

[Exclusion Criteria During Surgery] The patient who meets any criteria specified in the following 1) through 7).

1. Mechanical or surgical manipulation required to enlarge the pupil;
2. Excessive iris mobility;
3. Significant vitreous loss;
4. Significant anterior chamber hyphema;
5. Uncontrollable intraocular pressure;
6. Zonular or capsular rupture or tear;
7. IOL could not be fixed in the lens capsule;

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Binocular Best corrected distance visual acuity (5 m) | Postoperative Day 120-180 (4-6 months)
  CDVA measured with ETDRS charts placed in 5m distance with best aided corrective glasses according to ISO 11979-7:2014.
Binocular Distance corrected near visual acuity (40 cm) | Postoperative Day 120-180 (4-6 months)
  DCIVA measured with ETDRS charts placed in 40cm distance with corrective glasses for far distance according to ISO 11979-7:2014.
Binocular Distance corrected intermediate visual acuity (80 cm) | Postoperative Day 120-180 (4-6 months)
  DCIVA measured with ETDRS charts placed in 80cm distance with corrective glasses for far distance according to ISO 11979-7:2014.

SECONDARY OUTCOMES:
Binocular photopic best corrected distance visual acuity (5 m) | Postoperative Day 120-180
  DCIVA outcomes at 5m distance
Monocular and binocular photopic uncorrected distance visual acuity (5 m) | Postoperative Day 120-180
  UDVA outcomes at n 5m distance
Monocular and binocular photopic uncorrected intermediate visual acuity and binocular distance corrected intermediate visual acuity (80 cm) | Postoperative Day 120-180
  DCIVA outcomes at 80cm distance
Monocular and binocular photopic uncorrected near visual acuity and binocular distance corrected visual acuity (40cm) | Postoperative Day 120-180
  DCNVA outcomes at 40cm distance
Binocular photopic defocus curves | Postoperative Day 120-180
  To assess the visual acuity for different distances, defocus curves under photopic light conditions are measured. This test is performed with best distance corrected refraction and spherical additions ranging from -5.0 D to +1.5 D.
Contrast Sensitivity under photopic light conditions | Postoperative Day 120-180
  Contrast Sensitivity outcomes under photopic light conditions
Contrast Sensitivity under mesopic light conditions | Postoperative Day 120-180
  Contrast Sensitivity outcomes under photopic light conditions
Quality of Vison: VFQ-11 Questionnaire | Postoperative Day 120-180
  Outcomes measures of a questionnaire to address the general patient satisfaction and possible side effects of the treatment. For this study, the validated and verified Visual Functioning Questionnaire - 25 (VFQ-25) will be used. The maximum score for each questionaire is 100.

CONTACTS AND LOCATIONS:
Overall Officials: Kazunori Miyata, MD, PhD, Principal Investigator — Miyata Eye Hospital
Locations (1):
- Miyata Eye Hospital, Miyata, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mori Y, Miyata K, Suzuki H, Noguchi S, Ichikawa K, Maeda N. Clinical Performance of a Hydrophobic Acrylic Diffractive Trifocal Intraocular Lens in a Japanese Population. Ophthalmol Ther. 2023 Apr;12(2):867-878. doi: 10.1007/s40123-022-00634-4. Epub 2022 Dec 21. PMID 36542257
- [Derived] Mori Y, Miyata K, Kojima T, Ichikawa K, Fujita Y, Shiba T, Bissen-Miyajima H. Clinical performance of a hydrophobic acrylic toric intraocular lens with a double C-loop haptics in Japanese patients. Jpn J Ophthalmol. 2025 Sep 29. doi: 10.1007/s10384-025-01274-4. Online ahead of print. PMID 41021165
- See also: Official study publication of Clinical results — https://pubmed.ncbi.nlm.nih.gov/36542257/